CLINICAL TRIAL: NCT02185001
Title: Repair of Medial Patellofemoral Ligament Compared to Conservative Treatment for First Time Patella Dislocation; A Randomized Prospective Trial
Brief Title: Repair of Medial Patellofemoral Ligament Compared to Conservative Treatment for First Time Patella Dislocation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate patient recruitment and coordinator left organization
Sponsor: Orthopedic Specialty Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLKC-0001
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Dislocated Patella; Torn Medial Patellofemoral Ligament
Keywords: Medial patellofemoral ligament; MPFL; Repair; Patellar dislocation; Knee
MeSH Terms: conditions — Patellar Dislocation | interventions — Wound Healing; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical Treatment Group (Active Comparator): Direct Medial Patellofemoral Ligament (MPFL) Repair
  Interventions: Procedure: Direct Medial Patellofemoral Ligament (MPFL) Repair
- Conservative Treatment Group (Active Comparator): Immobilization, stabilization bracing, and physical therapy
  Interventions: Procedure: Physical therapy

INTERVENTIONS:
Procedure: Direct Medial Patellofemoral Ligament (MPFL) Repair — The MPFL will be repaired directly at the site of the traumatic injury.
  Other Names: Surgical Treatment Group
  Arms: Surgical Treatment Group
Procedure: Physical therapy — Patellar immobilization, stabilization, and strengthening under the direction and guidance of the physician and physical therapist.
  Other Names: Physiotherapy
  Arms: Conservative Treatment Group

SUMMARY:
Background: The forces involved in a patella dislocation event can cause significant collateral damage involving the articular cartilage of the patella femoral joint. As a result, prevention of recurrent patella dislocation and the associated disability and morbidity has generated significant interest in the orthopedic community. Historically, nonoperative treatment for first time patella dislocation has been problematic due to high redislocation rates. Nonoperative protocols generally involve bracing and/or immobilization, followed by physical therapy (1). Surgical approaches to recurrent patella dislocation, both soft tissue and boney realignment operations, have also had mixed results, including low success rates, associated complications, and variable rates of return to functional activity (2,3,4). This study is intended to compare the outcomes of a relatively low-risk Medial Patellofemoral Ligament (MPFL) direct repair procedure to conservative treatment.

Methods/Design: This study is designed as a two arm randomized prospective trial. Approximately fifty subjects will be randomly assigned to either a surgical or non-operative arm by means of a computer randomized allocation program. All subjects will have X-Ray Images and Magnetic Resonance Imaging (MRI) to determine the site of the MPFL damage, and to determine if any excluding conditions exist. Subjects randomized to the surgical group will have repair of the MPFL. Routine aftercare will consist of physical therapy in a clinic that has agreed to follow our protocol. Subjects randomized to the nonoperative group will receive 2 weeks of patellar immobilization, followed by patellar stabilization bracing with physical therapy for approximately 12 weeks. Physical therapy will progress through five phases with the goal of gait normalization, full range of motion and return to sport. Both arms will be given outcome questionnaires and physical activity assessments before treatment, and at one, three, six, twelve, and twenty four month intervals.

Discussion: This prospective randomized trial will investigate the results of direct repair of the medial patellofemoral ligament and conservative treatment by applying subjective outcome measures (Kujala scores), and exam findings to determine MPFL functional restoration or redislocation. Subjects will be examined in the clinic setting at 10 days, one month, and six months post trauma. Any reported recurrent dislocation or subluxation event will be documented during recovery. All subjects will receive merchant x-ray views at 3 months with manual lateral translation of the patella.

DETAILED DESCRIPTION:
Background Historic treatment for first time patella dislocation has been largely conservative. Treatment options include nonoperative treatment and a large variety of operative options. Nonoperative treatment, usually consists of bracing and/or immobilization followed by physical therapy, has been problematic due to a relatively high reported redislocation rate(1). The forces involved in a patella dislocation event can damage the articular cartilage of the patella femoral joint. As a result, prevention of recurrent patella dislocation and the associated disability and morbidity has generated significant interest in the orthopedic community.

Historic surgical approaches to recurrent patella dislocation have had mixed results. The isolated "lateral release", has been shown to have a very low success rate(2), while associated complications have been appreciated. Lateral release procedures are now more often performed in conjunction with other proximal or distal realignment procedures(3). More aggressive bone realignment procedures such as tibial tubercle transfers have the disadvantage of reported poor long term functional recoveries and low "return to sport" rates(4,5).

There has been increasing interest in ligament reconstruction for patella dislocation. The ligament of interest is the medial patella-femoral ligament (MPFL), which is essentially a thickened band of the medial capsule of the knee. The MPFL has been established as the primary constraint to patella dislocation. This ligament extends from a point just anterior to the attachment of the medial collateral ligament to the medial aspect of the patella, and is routinely disrupted with a patella dislocation event. The goals of reconstruction procedures are to replace and/or augment this band of tissue. While many reports of the results of MPFL reconstruction have been good to excellent, there are significant associated risks of complication, prolonged recovery, and associated graft costs or autograft harvest morbidity.

An alternative approach to MPFL functional restoration, and the subject of this study proposal, is a direct repair of the MPFL. Variations of this approach have been previously studied. A basic understanding of established injury patterns to the MPFL is requisite to evaluating the limitations to these studies.

Studies evaluating MPFL injury by MRI have shown that acute patella dislocations have a very high incidence of associated MPFL injury. The location of the lesion in the ligament can be described in one of four ways: 1) at the patellar attachment, 2) at the femoral attachment, 3) intrasubstance portion of the ligament, or 4) a combined injury pattern. Several studies have demonstrated varying percent distributions of injury(6,7), but it is clear that all patterns exist. This conclusion is consistent with the author's experience is treating these injuries.

Detecting the injury location can also be a challenge. Arthroscopic examination has been shown to be ineffective at determining the location of injury(8) and, in the experience of the author, MRI evaluation is frequently inaccurate, especially in the chronic or recurrent patella dislocation setting. The author proposes a functional intraoperative test to determine the ligament injury location.

Some prior reports have included surgical treatment of MPFL injuries using one technique only, with results similar to nonoperative treatment. For instance, some studies have evaluated treating all patella dislocations with repair at the patellar insertion, a treatment which may have limited or no benefit for patients with injuries at the femoral attachment of the ligament. There are two limited reports evaluating somewhat similar techniques, and these reports indicate some of the best results in the literature in the management of patella-femoral instability (9,10). These results are consistent with the author's experience with the treatment of this condition.

The subject of this study is to determine the difference in nonoperative and surgical patient outcomes using contemporary surgical techniques; identifying the location of the injury and choosing either direct repair or appropriate advancement. We hypothesize that minimally invasive surgical repair of the MPFL will improve patient outcomes and minimize recurrent patellar dislocation, when compared to conservative treatment. Our null hypothesis is that there will be no difference in outcomes between the two groups.

Methods/Design Trial Design - The study design will be a prospective parallel-group, randomized trial with allocation concealment.

Participants - At least 50 subjects will be recruited by referral from primary care providers, specialists, urgent care and emergency departments, and physical therapy clinics within a 50 mile radius of the clinic. Men, women, and minors, aged 10-17 will be recruited.

Inclusion criteria:

* A first patellofemoral traumatic dislocation
* A need for reduction
* An absence of fractures on x-ray exam of the frontal and lateral knee and axial patella
* An absence of knee ligament lesions with surgical indications (with the exception of the MPFL)
* No previous knee surgery

Exclusion criteria:

* A prior episode of patellofemoral dislocation
* Fractures on x-ray exam of the frontal and lateral knee and axial patella Prior surgery on the knee
* Tibial tuberosity-trochlear groove distance greater than 20mm
* Current pregnancy or plan to become pregnant during the study period. Recruitment - The recruitment process will consist of two phases. Phase one will consist of a short screening questionnaire, and phase two will consist of a clinical examination and questionnaire. Recruitment will remain open until at least fifty subjects that meet the inclusion criteria agree to participate.

Randomization - After screening and accepting subjects in the recruiting process, subjects will be randomly assigned to either an operative group or non-operative group by means of computer randomized sequencing and blind allocation. Random sequence generation will be done by using Random Allocation Software 1.0.0., and allocation will be concealed by placing allocations in sequentially numbered, sealed envelopes. Randomization, allocation, and concealment will be accomplished by an administrative assistant with no interest in the study or its outcome.

Interventions - All subjects will be briefed on their respective treatment protocols. The operative group will be advised on the risks of this surgery, including the chance of recurrent dislocations, as well as the more general risks of infection, DVT/PE, anesthesia complications, and associated possible complications (Table 1.1). The non-operative group will be advised of the possible failure of treatment, possibility of recurrent dislocation, and the possible need for surgery (Table 1.2).

All subjects will receive long standing and sunrise x-rays for diagnostic purposes. An MRI will be obtained for identifying the site of the lesion for both groups. Additionally, we will ask the subjects to complete a Kujala Scoring questionnaire and physical activity assessment as a baseline measurement, with the intention of evaluating and subjectively comparing the two types of treatment. Treatment for the surgical group will be performed at an outpatient surgical facility, and the non-operative group will receive treatment at a physical therapy clinic of their choice.

Surgical Treatment Group - Subjects who are randomized to the surgical group treatment will undergo surgical repair of their medial patellofemoral ligament. This will be identified using an MRI scan for the site of the lesion. If this cannot be identified, the following process will be used to determine the site of the lesion: On physical examination, the point of maximal tenderness between the patella and the femur will be identified and that will be the assumed site of traumatic injury to the medial patellofemoral ligament.

Surgery will be performed initially with a diagnostic arthroscopy to evaluate for loose bodies or chondral damage anywhere in the patellofemoral joint. A video will be taken of this and provided to the patient postoperatively. If there are no loose bodies or chondral damage to be treated, the medial patellofemoral ligament will then be repaired.

An incision will be made approximately 2 cm in length over the assumed site of the injury. The medial patellofemoral ligament will be identified and a tag suture will be applied to it. Traction on the medial patellofemoral ligament at this location will confirm that this is the site of primary injury by determining whether there is a firm endpoint with traction. If there is not a firm endpoint, a secondary incision over the alternate location, either the patella or the femur, will be made and the medial patellofemoral ligament will be identified in that location.

Repairs of the medial patellofemoral ligament will be made at all sites opened surgically whether it be either the femur or the patella, or both. Surgical repair will consist of providing decortication of the bone at the anatomic location of the medial patellofemoral ligament. Placement of a single 5 mm metal suture anchor with FiberWire-type sutures and a repair of the medial patellofemoral ligament using the FiberWire sutures to dock the ligament into its anatomic location. The repairs will be then be oversewn with #1 Vicryl suture at the site of the repair.

Following this, the local anesthetic will be applied to the incisions. They will be copiously irrigated and repaired with absorbable sutures.

The subjects will be placed in a hinged knee brace postoperatively with a range of motion restriction of 0-45 degrees. Weight bearing will be allowed immediately following surgery.

The subjects will start physical therapy the week of surgery and will begin with quadriceps strengthening with a restriction of range of motion from 0-45 for the first four weeks postoperatively followed by unrestricted full range of motion after week six. Full sport activities will be allowed to be resumed after eight weeks, provided the patient have at least 85% of the strength in their quadriceps compared to the contralateral side. Actual progression will be individualized based upon the patient's weekly reassessment and the presence of any complications.

Postoperative follow-ups will be made at the below-mentioned intervals with appropriate Kujala scoring and physical activity assessment (Table 2). X-rays will be taken on the first postoperative visit to confirm location of suture anchor repairs.

Appointments for physical examinations will be made at 7-10 days, 1 month, and three months after surgery. Any reported recurrent dislocation or subluxation event will be documented during recovery. All subjects will receive sunrise x-ray views at 3 months with manual lateral translation of the patella, as part of the study.

Conservative Treatment Group - The conservative treatment protocol is based on accepted physical therapy models of care and is established relative to patient tolerance for tissue healing, recovery, and response to modalities and procedures. Actual progression will be individualized based upon the patient's weekly reassessment and the presence of any complications. Prevention and minimization of recurrent dislocation, painful subluxation and osteoarthrosis are paramount in early management scenarios. The post traumatic and post surgical sequelae of pain, inflammation, swelling, bruising and muscular deactivation will be managed with acceptable standards of practice and prescribed medications. Prevention and dissipation of these sequelae, including modifying activities that put excessive stress or loading on the patellofemoral joint are the initial goals of rehabilitation in concert with gradual progression of mobility and muscular reactivation techniques. The protocol is divided into five phases: Phase I and II, 0-4 weeks; Phase III, 5-8 weeks; Phase IV- 9-12 weeks, Phase V- 13+ weeks (Table 3).

In addition to physical therapy appointments, subjects in the conservative treatment group will be given physical examination appointments and Kujala outcome scoring questionnaires and physical activity assessments at the same intervals as the surgical intervention group (Table 2). All subjects will receive sunrise x-ray views at 3 months with manual lateral translation of the patella, as part of the study.

Blinding-Due to the nature of the study, blinding of subjects after assignment to treatment groups is not feasible. All records and data will be collected and securely stored in the Clinical Research Coordinator's office. The data will be blinded before final statistical analysis by an independent statistician.

ELIGIBILITY:
Inclusion criteria:

* A first patellofemoral traumatic dislocation
* A need for reduction
* An absence of fractures on x-ray exam of the frontal and lateral knee and axial patella
* An absence of knee ligament lesions with surgical indications (with the exception of the MPFL)
* No previous knee surgery

Exclusion criteria:

* A prior episode of patellofemoral dislocation
* Fractures on x-ray exam of the frontal and lateral knee and axial patella Prior surgery on the knee
* Tibial tuberosity-trochlear groove distance greater than 20mm
* Current pregnancy or plan to become pregnant during the study period.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Patient Reported Change in Patellar Stability, Subluxation, or Recurrent Dislocation. | 24 months, or as reported by subject
  Subjects will be divided into 3 groups relating to patellar stability:
  1. Recurrence, indicating that the patient had a recurrent patellofemoral dislocation (total loss of congruence between the patella and trochlea) prior to 24 months.
  2. Unstable, indicating that the patient's knee presented with a positive apprehension test or showed signs of subluxation prior to 24 months, but without recurrent dislocation.
  3. Stable, indicating that the patient's knee did not show positive signs of episodes of subluxation at 24 months.

SECONDARY OUTCOMES:
Subjective Outcome Measurement (Kujala Test) | 1, 3, 6, 12, and 24 months
  Patients will be asked to complete the Kujala knee pain questionnaire to record pain and function levels at various points in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Lyman, MD, Principal Investigator — Orthopedic Specialty Institute
Locations (1):
- The Lyman Knee Clinic, Coeur d'Alene, Idaho, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maenpaa H, Huhtala H, Lehto MU. Recurrence after patellar dislocation. Redislocation in 37/75 patients followed for 6-24 years. Acta Orthop Scand. 1997 Oct;68(5):424-6. doi: 10.3109/17453679708996255. PMID 9385239
- [Background] Colvin AC, West RV. Patellar instability. J Bone Joint Surg Am. 2008 Dec;90(12):2751-62. doi: 10.2106/JBJS.H.00211. PMID 19047722
- [Background] Arendt EA, Fithian DC, Cohen E. Current concepts of lateral patella dislocation. Clin Sports Med. 2002 Jul;21(3):499-519. doi: 10.1016/s0278-5919(02)00031-5. PMID 12365240
- [Background] Arnbjornsson A, Egund N, Rydling O, Stockerup R, Ryd L. The natural history of recurrent dislocation of the patella. Long-term results of conservative and operative treatment. J Bone Joint Surg Br. 1992 Jan;74(1):140-2. doi: 10.1302/0301-620X.74B1.1732244.
- [Background] Aglietti P, Buzzi R, De Biase P, Giron F. Surgical treatment of recurrent dislocation of the patella. Clin Orthop Relat Res. 1994 Nov;(308):8-17. PMID 7955706
- [Background] Sillanpaa PJ, Peltola E, Mattila VM, Kiuru M, Visuri T, Pihlajamaki H. Femoral avulsion of the medial patellofemoral ligament after primary traumatic patellar dislocation predicts subsequent instability in men: a mean 7-year nonoperative follow-up study. Am J Sports Med. 2009 Aug;37(8):1513-21. doi: 10.1177/0363546509333010. Epub 2009 Apr 17. PMID 19376939
- [Background] Guerrero P, Li X, Patel K, Brown M, Busconi B. Medial patellofemoral ligament injury patterns and associated pathology in lateral patella dislocation: an MRI study. Sports Med Arthrosc Rehabil Ther Technol. 2009 Jul 30;1(1):17. doi: 10.1186/1758-2555-1-17. PMID 19643022
- [Background] Balcarek P, Walde TA, Frosch S, Schuttrumpf JP, Wachowski MM, Sturmer KM. MRI but not arthroscopy accurately diagnoses femoral MPFL injury in first-time patellar dislocations. Knee Surg Sports Traumatol Arthrosc. 2012 Aug;20(8):1575-80. doi: 10.1007/s00167-011-1775-7. Epub 2011 Nov 18. PMID 22095485
- [Background] Tom A, Fulkerson JP. Restoration of native medial patellofemoral ligament support after patella dislocation. Sports Med Arthrosc Rev. 2007 Jun;15(2):68-71. doi: 10.1097/JSA.0b013e31803035d3. PMID 17505320
- [Background] Camanho GL, Viegas Ade C, Bitar AC, Demange MK, Hernandez AJ. Conservative versus surgical treatment for repair of the medial patellofemoral ligament in acute dislocations of the patella. Arthroscopy. 2009 Jun;25(6):620-5. doi: 10.1016/j.arthro.2008.12.005. Epub 2009 Feb 26. PMID 19501292